CLINICAL TRIAL: NCT03246009
Title: Efficacy and Safety Phase Ib Study of Recombinant Human Serum Albumin/ Granulocyte Colony-Stimulating Factor Fusion Protein for Injection to Prevent Neutrophilic Granulocytopenia Among Chemotherapy Patients
Brief Title: Fusion Protein rHSA/GCSFclinical Study on Breast Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tianjin SinoBiotech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG01N-1399
Record Dates: First submitted 2017-08-08; First posted 2017-08-10 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Chemotherapy-induced Neutropenia; Cancer, Breast
Keywords: Neutropenia; Chemotherapy; rHSA/GCSF
MeSH Terms: conditions — Breast Neoplasms; Neutropenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- single injection-1.8mg (Experimental): rHSA/GCSF,injection,1.8mg,Single subcutaneous injection,Duration 1 day
  Interventions: Drug: rHSA/GCSF
- single injection-2.1mg (Experimental): rHSA/GCSF,injection,2.1mg,Single subcutaneous injection,Duration 1 day
  Interventions: Drug: rHSA/GCSF
- single injection-2.4mg (Experimental): rHSA/GCSF,injection,2.4mg,Single subcutaneous injection,Duration 1 day
  Interventions: Drug: rHSA/GCSF
- multiple injection-1.8mg (Experimental): rHSA/GCSF,injection,1.8mg, subcutaneous injection,Duration 4 day,A total of 2 injections, each interval of 3 days.
  Interventions: Drug: rHSA/GCSF
- multiple injection-2.1mg (Experimental): rHSA/GCSF,injection,2.1mg, subcutaneous injection,Duration 4 day,A total of 2 injections, each interval of 3 days.
  Interventions: Drug: rHSA/GCSF
- multiple injection-2.4mg (Experimental): rHSA/GCSF,injection,2.4mg, subcutaneous injection,Duration 4 day,A total of 2 injections, each interval of 3 days.
  Interventions: Drug: rHSA/GCSF

INTERVENTIONS:
Drug: rHSA/GCSF — single injection-1.8mg
  Arms: single injection-1.8mg
Drug: rHSA/GCSF — single injection-2.1mg
  Arms: single injection-2.1mg
Drug: rHSA/GCSF — single injection-2.4mg
  Arms: single injection-2.4mg
Drug: rHSA/GCSF — multiple injection-1.8mg
  Arms: multiple injection-1.8mg
Drug: rHSA/GCSF — multiple injection-2.1mg
  Arms: multiple injection-2.1mg
Drug: rHSA/GCSF — multiple injection-2.4mg
  Arms: multiple injection-2.4mg

SUMMARY:
The purpose of this study is to evaluate the tolerance and safety of the rHSA/GCSF in breast cancer patients with different doses and multiple injections.

To observe the pharmacokinetic characteristics of recombinant human serum albumin /granulocyte colony-stimulating factor fusion protein after single and multiple administration

DETAILED DESCRIPTION:
This experiment adopts the method of multicenter, open, dose escalation study injection with recombinant human blood clean protein/granulocyte stimulating factor fusion protein after single and multiple doses of tolerance, security, and pharmacokinetic characteristics.

Breast cancer patients with reduced white blood cells after chemotherapy were selected as subjects of this study.

The three research doses that were to be incremented were 1.8 mg, 2.1mg and 2.4mg respectively, each of which was studied by single and multiple doses.

Single dose of medicine, dose-climbing study.Two doses of the drug, dose-climbing study

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65.
* Diagnosed breast cancer，received chemotherapy.
* ECOG performance status 0 or 1.
* ANC≥1.5×10 9/L, PLT≥100×10 9/L. No bone marrow metastasis,blood coagulation function normally, no Hemorrhagic tendency.
* Leukocyte reduction occurred after chemotherapy,WBC≤3.0x109/L or ANC≤1.5x109/L.
* No obvious abnormal ecg examination.
* Cr，TBIL, AST, ALT≤1.5×ULN，no serious underlying disease.
* Signed informed consent.

Exclusion Criteria:

* Chemotherapy within past 4 weeks.
* Uncontrolled inflammatory disease,axillary temperature≥38℃.
* Merging other malignant tumor.
* Pregnancy or nursing status.
* Participation in another clinical trial with and investigational product within 3 months prior to study entry.
* Severe diabetes mellitus, or poor blood sugar controller.
* Allergic disease or allergic constitution. History of protein allergy.
* History of drug addiction and alcoholism.
* Hematopoietic stem cell transplantation or organ transplantation.
* Received antibiotic treatment within 72 hours before chemotherapy.
* Long-term use of hormones or immunosuppressive agents.
* Severe mental or neurological disorders.
* Chronic disease of severe cardiac, kidney and liver.
* Other conditions that would be excluded from this study according to doctors'judgment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-01-21 (Actual); Primary Completion 2017-04-10 (Actual); Study Completion 2017-04-10 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | 14 days
  Number of participants with AE as a measure for safety and tolerability after single and multiple dose of rHSA/GCSF

SECONDARY OUTCOMES:
AUC | 14 days
  AUC after single and multiple dose of rHSA/GCSF

CONTACTS AND LOCATIONS:
Overall Officials: Binghe XU, MD, Principal Investigator — chinese academy of medical sciences tumor hospital
Locations (1):
- Chinese Academy of Medical Sciences Cancer Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Chen S, Han Y, Ouyang Q, Lu J, Zhang Q, Yang S, Wang J, Huang H, Liu H, Shao Z, Li H, Chen Z, Sun S, Geng C, Lu J, Sun J, Wang J, Xu B. Randomized and dose-escalation trials of recombinant human serum albumin /granulocyte colony-stimulating factor in patients with breast cancer receiving anthracycline-containing chemotherapy. BMC Cancer. 2021 Mar 31;21(1):341. doi: 10.1186/s12885-021-08093-z. PMID 33789616